CLINICAL TRIAL: NCT02902107
Title: A Pilot Feasibility Trial of Unidirectional Low Dose Rate Brachytherapy for Patients With Abdominal and Pelvic Malignancy Undergoing Surgical Resection Requiring Intraoperative Radiation Therapy
Brief Title: Intraoperative Radiation Therapy for Locally Advanced or Recurrent Abdomino-pelvic Solid Tumors With the CivaSheet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: CivaTech Oncology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-605
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Abdominal Malignancy; Pelvic Malignancy
Keywords: Low Dose Rate Brachytherapy; CivaSheet; 16-605
MeSH Terms: interventions — Brachytherapy

ARMS (1):
- surgical resection and intraoperative radiation therapy (IORT) (Experimental): Brachytherapy will be administered using the CivaSheet, a novel permanent LDR palladium-103 (Pd-103) planar brachytherapy device that is applied directly to the surgical resection bed.
  Interventions: Device: CivaSheet; Radiation: Brachytherapy; Procedure: surgical resection

INTERVENTIONS:
Device: CivaSheet
Radiation: Brachytherapy
Procedure: surgical resection

SUMMARY:
This study is a pilot study of the CivaSheet, a new type of intraoperative radiation therapy (IORT) device that offers several advantages over existing techniques of performing IORT. The CivaSheet device in this study is already approved by the FDA and is not an experimental device. This study will allow us to determine how feasible it is to implant the CivaSheet into patients undergoing surgery for abdominal and pelvic tumors, and assess any possible side effects of the device. This study, if successful, may allow us to offer the CivaSheet more widely as treatment option to future patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologic, cytologic, or radiologically evidence of locally advanced, residual or recurrent solid malignancy of the abdomen or pelvis requiring surgical resection
* Maximum projected treatment length 15cm and width 5cm, which are the dimensions of the largest available CivaSheet
* Medically fit and willing to undergo resection of disease
* Age ≥ 18 years
* ECOG performance status 0, 1, or 2
* ANC ≥ 1.5 cells/mm3, PLT≥100,000/mm3, PT/aPTT within normal limits at time of surgery
* Life expectancy, in the clinician's judgment, greater than 1 year.

Exclusion Criteria:

* Women who are pregnant
* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy after the receipt of brachytherapy. Male subjects must also agree to use effective contraception during the treatment period and until 1 year after the completion of brachytherapy
* Patients with any concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study.
* Patients who, in the investigator's judgment, are unwilling or unable to consent to and return for recommended post-treatment scans as outlined in this study.
* Patients on concurrent anti-cancer therapy, unless specifically agreed to by the patient's medical oncologist and consenting professional.
* Patients with contraindications to general anesthesia, as determined by the treating physician or surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2016-09-09 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
number of successful implantation of the device in patients | 1 year
  Feasibility is determined by successful implantation of the device into a patient who has been enrolled on the protocol and deemed appropriate for IORT at the time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Wu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/